CLINICAL TRIAL: NCT05609487
Title: Evaluation of the Effectiveness of the Implementation of a Safety Plan by the Emergency Nurse to Prevent Suicidal Reiteration - National Multicenter Randomized Controlled Trial in Stepped-wedge
Brief Title: Evaluation of the Safety Plan to Prevent Suicidal Reiteration
Acronym: PROTECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2022-A00163-40
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Suicide, Attempted
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: The study is structured in three phases: 1) translation and adaptation of the safety plan into French; 2) effectiveness study; and 3) evaluation of the implementation of the safety plan in practice
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Step in "control group" This stepped wedge study does not use two parallel treatment arms. The stepped wedge design allows each center to be its own "control group" and then, after implementation of the practice by the research team, to become a "intervention group".
  The characteristics of these two phases are detailed below. Patients included in the control phase, i.e. without intervention, will be asked not to oppose participation in the research, after having received the presentation of the study and the information notice. The data collection will be similar to the data collection during the intervention period.
  Interventions: Other: As usual
- Protection plan group (Other): The intervention consists of making the protection plan in a co-constructed process with the care user. This tool is built in 6 steps, is written and takes 20 to 40 minutes to complete.
  These 6 steps allow to identify the first signs of a suicidal crisis and to identify different strategies to face it. They are constructed in an ascending order, with the aim of being used by the care user in an autonomous situation.
  Interventions: Device: Protection plan

INTERVENTIONS:
Other: As usual — Patients included in the control phase, i.e. without intervention, will be asked not to oppose participation in the research, after having received the presentation of the study and the information notice. The data collection will be similar to the data collection during the intervention period.
  Arms: Control group
Device: Protection plan — The intervention consists of making the protection plan in a co-constructed process with the care user. This tool is built in 6 steps, is written and takes 20 to 40 minutes to complete.
  These 6 steps allow to identify the first signs of a suicidal crisis and to identify different strategies to face it. They are constructed in an ascending order, with the aim of being used by the care user in an autonomous situation.
  Arms: Protection plan group

SUMMARY:
Each year, suicide is the cause of 8,580 deaths in France, it is the second leading cause of death among 15-24 year olds. People who have made a first suicide attempt are identified as being at greater risk of repeating a suicidal gesture, particularly in the first month following the gesture . At the same time, Brief Intervention Contact (BIC) is recognized as effective in reducing suicide deaths.

A new brief intervention to prevent suicidal attempts has been developed in the United States by Santley & Brown (2012) the results of its effectiveness are very encouraging.

Investigators hypothesise that the implementation of a safety plan by the emergency department for suicidal patients included in the Vigilans system leads to a greater reduction in the reiteration of suicidality at 6 months compared to the usual management.

Our main objective is to evaluate the effectiveness of the implementation of a safety plan by the emergency department nurse before discharge from the emergency department in reducing suicidal reiteration at six months after the suicide attempt, for suicidal patients included in the Vigilans programe, compared with the Vigilans programe alone.

Our secondary objectives are

* Reduce the reiteration of the suicidal act at 1 month
* Encourage engagement in care at 1 month and 6 months
* Reduce the use of emergency departments at 1 month and 6 months due to a suicidal crisis
* Decrease suicide mortality at 6 months

To study the implementation of the intervention:

* To measure the quality of completion, and the duration of completion of the safety plan at 1 month, and 6 months.
* Assess the acceptability of the safety plan by emergency department nurses, and then by the vigilantes.
* Assess the acceptability of the safety plan by patient

DETAILED DESCRIPTION:
Each year, suicide is the cause of 8,580 deaths in France , and although the suicide rate in France has decreased by 10% over the last ten years, it is the second leading cause of death among 15-24 year olds.

People who have made a first suicide attempt are identified as being at greater risk of repeating a suicidal gesture, particularly in the first month following the gesture . At the same time, Brief Intervention Contact (BIC) is recognised as effective in reducing suicide deaths.

In 2012, two American psychiatrists developed and evaluated the effectiveness of a tool for preventing the recurrence of suicide: the safety plan. It consists of a list of strategies co-constructed by a trained health professional with the person concerned, which make it possible to deal with thoughts of suicide. It is deployed in 6 steps.

Once completed, it is kept by the user and can be used in complete autonomy at the first signs of a potential suicidal crisis.

This prevention tool, whose initial results across the Atlantic are very encouraging, is not used in daily practice in France.

The main objective of the study is therefore to evaluate its effectiveness at 6 months when it is implemented by the emergency room nurse, before discharge, for people already included in the VigilanS programme.

The VigilanS programme is the national system for preventing suicidal recurrence and consists of three complementary strategies:

1. Firstly, a resource card indicates a toll-free number, open during the day, for people who have made a gesture. Respondents are health professionals (vigilance workers) who can assess and guide people in the event of a recurrence of suicidal thoughts.
2. Then investigators contact the person's existing care network, investigators inform the attending doctor, but also other care providers (psychologist, physiotherapist, liberal nurse...) of their patient's inclusion in the system.
3. Finally, telephone calls are made by the health professionals in the first month following discharge, and six months after the suicidal act. In parallel, a postcard is sent monthly during the first 4 months to continue the link.

This national study will work with 11 hospitals with a Vigilans service and will be implemented in 19 emergency departments. Doctors, nurses and health managers will be identified in each center.

The first step of the study is to translate the tool (the safety plan), with the help of a committee of experts and specialized translators.

Then investigators will evaluate its effectiveness with 2,387 study participants included in the 19 emergency departments over a two-year period.

Each participating center (the emergency department) will initially be in an observation (or control) phase, i.e. the safety plan will not be used by the care workers. Then in a second phase, the research team will implement the practice of the tool through training, and in a third phase the center will be in the intervention phase, i.e. it will use the tool in daily practice.

The order of training, where the practice is implemented in the units, is chosen by randomization.

The main objective of the study is to evaluate six months after the suicide attempt, by a telephone call that will ask the patient if he or she has made a suicidal attempt again.

Investigators will thus be able to compare a population that has not received the tool (the control group) with a population that has received the tool (the intervention group) and thus measure its effectiveness.

Finally, the last stage of the study consists of evaluating the use of the tool by emergency service professionals, the Vigilans device, and the participants in the study. To do this, investigators will use questionnaires (evaluation scales) and conduct semi-structured interviews with several participants

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Seen in an emergency department
* Admitted in emergency department following a suicide attempt <48h
* whose duration of care does not exceed 24 hours
* For whom the care project results in a return home,
* Who agree to be included in the Vigilans system
* Who have social security coverage
* Fluent in French

Exclusion Criteria:

* Refusal to participate in the study
* Refusal to be accompanied by the Vigilans system
* Hospitalisation for more than 24 hours in the immediate aftermath of the suicide attempt
* Under protective measures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2387 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Suicidal recurrence at 6 months | 6 months
  Suicidal reiteration is characterized by non-fatal suicidal behavior, self-inflicted injury with a desire to end one's life that does not result in death (WHO).

SECONDARY OUTCOMES:
Suicidal recurrence | one month
  Suicidal reiteration is characterized by non-fatal suicidal behavior, self-inflicted injury with a desire to end one's life that does not result in death (WHO).
Commitment to healthcare | One month and 6 months
  Currently in mental health care? Y/N number of appointments in mental health care since the suicide attempt
Death by suicide attempt | 6 months
  Collected by cross-referencing information from the Vigilans system, by contacting the doctor or family members and other contacts. In the event of a lost person with no vital status data, civil status registers may be used.

CONTACTS AND LOCATIONS:
Overall Officials: BENOIT CHALANCON, IDE, Principal Investigator — CH LE VINATIER
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, AURA, France

REFERENCES:
- [Derived] Chalancon B, Haesebaert J, Vacher A, Vieux M, Simon L, Subtil F, Colin C, Poulet E, Leaune E; Investigator Associates; Expanded Scientific Nursing Committee. Implementing a nurse-led safety planning intervention in emergency departments to prevent suicide reattempts: a stepped-wedge randomized controlled trial protocol (French multicentre randomized controlled trial with a stepped-wedge design). BMC Nurs. 2025 May 19;24(1):558. doi: 10.1186/s12912-025-03121-w. PMID 40389942